CLINICAL TRIAL: NCT05378945
Title: A Phase 3, Multicenter, Randomized, Controlled, Double-Masked Clinical Trial to Evaluate the Efficacy and Safety of OC-01 (Varenicline Solution) Nasal Spray on Signs and Symptoms of Dry Eye Disease in Chinese Population
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of OC-01 (Varenicline) Nasal Spray on Signs and Symptoms of Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Corxel Pharmaceuticals (Industry)
Collaborators: Oyster Point Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JX03002
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Dry Eye Disease
Keywords: OC-01; Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- OC-01 (Experimental)
  Interventions: Drug: Varenicline Tartrate Nasal Spray
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (vehicle)

INTERVENTIONS:
Drug: Varenicline Tartrate Nasal Spray — Intranasal delivery of OC-01 (varenicline solution) 0.6 mg/mL twice a day (BID) for 28 days
  Other Names: OC-01 (varenicline solution) Nasal Spray
  Arms: OC-01
Drug: Placebo (vehicle) — Intranasal delivery of placebo (vehicle) twice a day (BID) for 28 days
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of OC-01 (varenicline solution) Nasal Spray as compared to placebo (vehicle) on signs and symptoms of dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Have used and/or desired to use an artificial tear substitute for dry eye symptoms within 6 months prior to the Screening Visit

Exclusion Criteria:

* Have had any intraocular surgery (such as cataract surgery) or extraocular surgery in either eye within three months or refractive surgery (e.g., laser-assisted in-situ keratomileusis, laser epithelial keratomileusis, photorefractive keratectomy or corneal implant) within 12 months of the Screening Visit
* Have a history or presence of any ocular disorder or condition in either eye that would, in the opinion of the Investigator, likely interfere with the interpretation of the study results or participant safety such as significant corneal or conjunctival scarring; pterygium or nodular pinguecula; current ocular infection, acute conjunctivitis, or inflammation not associated with dry eye; anterior (epithelial) basement membrane corneal dystrophy or other clinically significant corneal dystrophy or degeneration; ocular herpetic infection; evidence of keratoconus; etc. Blepharitis not requiring treatment and mild meibomian gland disease that are typically associated with DED are allowed.
* Have a systemic condition or disease not stabilized or judged by the Investigator to be incompatible with participation in the study (e.g., current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease, history of myocardial infarction or heart disease, etc.)
* Have a known hypersensitivity to any of the procedural agents or investigational product components
* Have any condition or history that, in the opinion of the investigator, may interfere with study compliance, outcome measures, safety parameters, and/or the general medical condition of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Schirmer's Test Score | 28 days
  Percentage of subjects who achieve ≥10 mm improvement in Schirmer's Test Score from baseline

SECONDARY OUTCOMES:
Mean change from Baseline in Schirmer's Test Score (STS) | 28 days
  Schirmer's test scores are from 0-35 mm where a higher score is indicative of a better outcome.
Mean change from Baseline in Eye Dryness Score (EDS) | 28 days/ 14 days/ 7days
  Eye dryness score is assessed on a visual analogue scale with scores ranging from 0 to 100 (0=no discomfort; 100=maximal discomfort) and lower scores indicate a better outcome

OTHER OUTCOMES:
Mean change from Baseline in Total Corneal Fluorescein Staining | 28 days
Mean change from Baseline in Inferior Corneal Fluorescein Staining | 28 days
Mean change from Baseline in Nasal Corneal Fluorescein Staining | 28 days
Mean change from Baseline in Temporal Corneal Fluorescein Staining | 28 days
Mean change from Baseline in Central Corneal Fluorescein Staining | 28 days
Mean change from Baseline in Superior Corneal Fluorescein Staining | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: JIE, Doctor, Principal Investigator — Beijing Tongren Hospital; DING, Study Director — Corxel Pharmaceuticals
Locations (20):
- China (20):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Tongren Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Shijiazhuang People's Hospital, Shijiazhuang, Hebei
  - Hebei Eye Hospital, Xingtai, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Eye Hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Aier Eye Hospital Hankou Hospital, Wuhan, Hubei
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Eye Hospital of Shandong First Medical University, Jinan, Shandong
  - Weifang Eye Hospital, Weifang, Shandong
  - Shanghai Ninth People's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang